CLINICAL TRIAL: NCT03737968
Title: Window of Opportunity Trial of Durvalumab (MEDI4736) or Durvalumab/Tremelimumab as Neoadjuvant Chemotherapy to Identify Immune Dynamics in Surgically Resectable Head and Neck Cancer Patients.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2018-0787
Record Dates: First submitted 2018-11-08; First posted 2018-11-13 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Stage II-IVB Operable HNSCC Oral Cavity; Hypopharynx; Oropharynx; Larynx
Keywords: oral cavity; hypopharynx; oropharynx; larynx; medi4736; tremelimumab
MeSH Terms: conditions — Laryngeal Diseases | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Durvalumab monotherapy Arm (Experimental): Patients in the durvalumab (MEDI4736) monotherapy treatment group will receive durvalumab (MEDI4736) (1500mg Q4W) once prior to surgery in this study. After surgical resection, these patients will receive the post op adjuvant treatment including RTx with/without cisplatin based on the pathologic findings and physician's discretion. After completion of adjuvant treatment, durvalumab (MEDI4736) 1500mg Q4W as maintenance treatment for up to a maximum of 12 months until confirmed disease progression unless there is unacceptable toxicity, withdrawal of consent, or another discontinuation criterion is met. The first durvalumab (MEDI4736) monotherapy dose at 1500mg Q4W will be within 8 weeks after the completion of adjuvant therapy. If a patient's weight falls to 30kg or below the patient should receive weight-based dosing equivalent to 20 mg/kg of durvalumab Q4W until the weight improves to >30 kg, at which point the patient should start receiving the fixed dosing of durvalumab 1500mg.
  Interventions: Drug: Durvalumab
- Durvalumab + tremelimumab combination therapy Arm (Active Comparator): Patients in the durvalumab (MEDI4736) + tremelimumab combination therapy treatment group will receive durvalumab (MEDI4736) (1500mg Q4W) in combination with tremelimumab (75 mg IV Q4W) once prior to surgery in this study. After surgical resection, these patients will receive the post op adjuvant treatment including RTx with/without cisplatin based on the pathologic findings and physician's discretion. After completion of adjuvant treatment, durvalumab (MEDI4736) 1500mg Q4W as maintenance treatment for up to a maximum of 12 months until confirmed disease progression unless there is unacceptable toxicity, withdrawal of consent, or another discontinuation criterion is met. The first durvalumab (MEDI4736) monotherapy dose at 1500mg Q4W will be within 8 weeks after the completion of adjuvant therapy.
  Interventions: Drug: durvalumab + tremelimumab

INTERVENTIONS:
Drug: Durvalumab — Patients in the durvalumab (MEDI4736) monotherapy treatment group will receive durvalumab (MEDI4736) (1500mg Q4W) once prior to surgery in this study. After surgical resection, these patients will receive the post op adjuvant treatment including RTx with/without cisplatin based on the pathologic findings and physician's discretion. After completion of adjuvant treatment, durvalumab (MEDI4736) 1500mg Q4W as maintenance treatment for up to a maximum of 12 months
  Arms: Durvalumab monotherapy Arm
Drug: durvalumab + tremelimumab — Patients in the durvalumab (MEDI4736) + tremelimumab combination therapy treatment group will receive durvalumab (MEDI4736) (1500mg Q4W) in combination with tremelimumab (75 mg IV Q4W) once prior to surgery in this study. After surgical resection, these patients will receive the post op adjuvant treatment including RTx with/without cisplatin based on the pathologic findings and physician's discretion. After completion of adjuvant treatment, durvalumab (MEDI4736) 1500mg Q4W as maintenance treatment for up to a maximum of 12 months
  Arms: Durvalumab + tremelimumab combination therapy Arm

SUMMARY:
This is a phase II randomized, open label study of durvalumab with/ without tremelimumab as neoadjuvant therapy and durvalumab maintenance after SoC RTx with/without cisplatin as post-surgical adjuvant therapy in treatment naïve participants with newly diagnosed resectable LA HNSCC. The study will be conducted in conformance with Good Clinical Practices (GCP). Approximately 44 participants will be randomized in a 1:1 ratio to below two Arms

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed surgically resectable HNSCC oral cavity, hypopharynx, oropharynx, and larynx
* Measurable disease defined as lesions that can be accurately measured by RECIST 1.1.
* Written informed consent and any locally-required authorization obtained from the patient prior to performing any protocol-related procedures, including screening evaluations
* Age >18 years at time of study entry or Adult male or female
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Body weight >30kg
* Life expectancy of at least 12 weeks
* Adequate normal organ and marrow function as defined below:

  * Haemoglobin ≥9.0 g/dL
  * Absolute neutrophil count (ANC) > 1500 per mm3
  * Platelet count >75,000 per mm3
  * Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN).
  * AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤5x ULN
  * Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine clearance CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

Males: Creatinine CL (mL/min) = Weight (kg) x (140 - Age) 72 x serum creatinine (mg/dL) Females: Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL)

Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

* Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
* Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

Involvement in the planning and/or conduct of the study Participation in another clinical study with an investigational product during the last Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.

History of allogenic organ transplantation. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

* Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
* Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the Study Physician.

Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.

Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

* Patients with vitiligo or alopecia
* Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
* Any chronic skin condition that does not require systemic therapy
* Patients without active disease in the last 5 years may be included but only after consultation with the study physician
* Patients with celiac disease controlled by diet alone Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent History of another primary malignancy except for
* Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence
* Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
* Adequately treated carcinoma in situ without evidence of disease History of active primary immunodeficiency Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.

:Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or tremelimumab. The following are exceptions to this criterion:

* Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
* Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.

Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy or 180 days after the last dose of durvalumab + tremelimumab combination therapy.

Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.

Prior treatment with an anti-PD-1, anti-PD-L1 (including durvalumab), anti-PD-L2, anti-CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including tremelimumab).

Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 180 days after the last dose of durvalumab + tremelimumab combination therapy or 90 days after the last dose of durvalumab monotherapy, whichever is the longer time period

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
locoregional relapse rate | every 3 months, assessed up to 2 years
  investigate the locoregional relapse rate (LRR)
Distant metastatic rate | every 3 months, assessed up to 2 years
  Distant metastatic rate

SECONDARY OUTCOMES:
distant metastases free survival (DMFS) | every 3 months, assessed up to 2 years
locoregional control (LRC) time | every 3 months, assessed up to 2 years
progression-free survival (PFS) | every 3 months, assessed up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cha J, Kim CG, Sim NS, Kim G, Son W, Kim D, Jung Y, Hong HJ, Lee HB, Kim J, Kim J, Yoon SO, Go S, Kim J, Seong E, Baek S, Kim KH, Hong MH, Koh YW, Lee I, Kim HR. 4-1BB+ Tregs and inhibitory progenitor exhausted T cells confer resistance to anti-PD-L1 and anti-CTLA-4 combination therapy. Cell Rep Med. 2025 Oct 21;6(10):102408. doi: 10.1016/j.xcrm.2025.102408. Epub 2025 Oct 3. PMID 41045934
- [Derived] Cha J, Kim DH, Kim G, Cho JW, Sung E, Baek S, Hong MH, Kim CG, Sim NS, Hong HJ, Lee JE, Hemberg M, Park S, Yoon SO, Ha SJ, Koh YW, Kim HR, Lee I. Single-cell analysis reveals cellular and molecular factors counteracting HPV-positive oropharyngeal cancer immunotherapy outcomes. J Immunother Cancer. 2024 Jun 10;12(6):e008667. doi: 10.1136/jitc-2023-008667. PMID 38857913